CLINICAL TRIAL: NCT00501241
Title: A Phase II, Randomized, Placebo-Controlled Study of ATI-7505 in Patients With Chronic Idiopathic Constipation
Brief Title: Phase II, Randomized, Placebo-Controlled Study of ATI-7505 in Patients With Chronic Idiopathic Constipation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Tom Todaro, MD, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007003
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2008-02

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — ATI 7505

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): placebo twice daily
  Interventions: Drug: ATI-7505
- 2 (Experimental): 20 mg ATI-7505, BID for 4 weeks
  Interventions: Drug: ATI-7505
- 3 (Experimental): 40 mg ATI, BID, 4 weeks
  Interventions: Drug: ATI-7505
- 4 (Experimental): 80 mg ATI-4505, BID for 4 weeks
  Interventions: Drug: ATI-7505
- 5 (Experimental): 120 mg ATI-7505, BID for 4 weeks
  Interventions: Drug: ATI-7505

INTERVENTIONS:
Drug: ATI-7505 — Tablet,placebo, BID
  Arms: 1
Drug: ATI-7505 — ATI-7505 20 mg BID for 4 weeks
  Arms: 2
Drug: ATI-7505 — tablet, 40 mg, BID, $ weeks
  Arms: 3
Drug: ATI-7505 — 80 mg ATI-7505, BID for 4 weeks
  Arms: 4
Drug: ATI-7505 — 120 mg ATI-7505, BID, for 4 weeks
  Arms: 5

SUMMARY:
The purpose of this study is to determine whether ATI-7505 is effective in the treatment of chronic idiopathic constipation.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of ATI 7505 in generally healthy, adult patients who have had symptoms of chronic idiopathic constipation for at least 6 months as defined in the ROME III criteria.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* 18 and 75 years of age
* constipation symptom onset at least 6 months ago & meet ROME III criteria for chronic constipation
* negative colonoscopy or air contrast barium enema within the past 2 years if ≥50 years of age or within the past 5 years if <50 years of age;
* are able to refrain from use of medications known to treat constipation or associated symptoms throughout the study

Exclusion Criteria:

* transabdominal surgery, unstable coronary artery disease, organic gastrointestinal disease, collagen vascular disease, or any alarm symptoms within the 6 months prior to screening;
* taking prohibited medications (including laxatives, herbal remedies)
* participating in another drug or medical device study or use of any investigational drug within 30 days before dosing or planning to use prior to study completion;
* QTcB >440 msec, abnormal 12-lead ECG, family history of sudden death at age <40 years or history of long QT syndrome
* alcohol or drug abuse within the 6 months prior to screening;
* autonomic dyssynergic defecation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Total number of spontaneous bowel movements during the first 7 days after randomization | 7 days

SECONDARY OUTCOMES:
Daily and/or weekly assessments of the consistency, severity, frequency, symptoms of constipation during the treatment period | daily and or weekly

CONTACTS AND LOCATIONS:
Overall Officials: Tom G Todaro, MD, Study Director — Procter and Gamble
Locations (23):
- United States (20):
  - Research Facility, Anaheim, California
  - Research facility, San Carlos, California
  - Research Facility, San Diego, California
  - Research Facility, Littleton, Colorado
  - Research Facility, Aventura, Florida
  - Research Facility, Hollywood, Florida
  - Research Facility, South Miami, Florida
  - Researrch Facility, Newnan, Georgia
  - Research Facility, Rockford, Illinois
  - Research Facility, Evansville, Indiana
  - Research Facility, Boston, Massachusetts
  - Research Facility, Great Neck, New York
  - Research Facility, Lake Success, New York
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Oklahoma City, Oklahoma
  - Research Facility, Chattanooga, Tennessee
  - Research Facility, Nashville, Tennessee
  - Research Facility, Salt Lake City, Utah
  - Research Facility, Charlottesville, Virginia
  - Research Facility, Christiansburg, Virginia
- Canada (3):
  - Research Facility, Montreal, Quebec
  - Reserach Facility, Québec, Quebec
  - Research Facility, Saint Charles Borremee, Quebec